CLINICAL TRIAL: NCT02782156
Title: Evaluation of the Standardised Nurse-led Approach for Risk Screening and Decrease of Alcohol Withdrawal Among Adult Inpatients With Alcohol Dependence in an Ear, Nose, Throat and Jaw Surgery Department
Brief Title: Process Evaluation Standardised Nurse-led Approach for Risk Screening and Decrease of Alcohol Withdrawal in ENT
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2014-318
Record Dates: First submitted 2015-06-15; First posted 2016-05-25 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Substance Withdrawal Syndrome
Keywords: Process Evaluation; alcohol withdrawal syndrome
MeSH Terms: conditions — Substance Withdrawal Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Process evaluation — Adherence to screening and action algorithm

SUMMARY:
In ear, nose, throat (ENT) and jaw surgery departments, up to 60% of patients suffer from alcohol dependence (Allen et al., 2009), and may develop an alcohol withdrawal syndrome (AWS) when undergoing sur-gery. Caring for these patients creates a major challenge for all persons involved: Health care staff is not only challenged by the primary illness but also by increased risk of life-threatening complications (infection, bleeding, cardiopulmonary dysfunction, impaired wound healing, re-operation), higher mortality rate, and longer duration of hospitalization due to preoperative alcohol use and the development of an AWS (Delgado-Rodriguez, Gomez-Ortega, Mariscal-Ortiz, Palma-Perez, & Sillero-Arenas, 2003; Eyer et al., 2011; Foy, Kay, & Taylor, 1997; Genther & Gourin, 2012; Kuo et al., 2008; Mayo-Smith et al., 2004; McCusker, Cole, Abrahamowicz, Primeau, & Belzile, 2002; Neyman, Gourin, & Terris, 2005; O'Brien et al., 2007). Moreover, nearly five percent of all patients with an AWS develop an alcohol withdrawal delirium (AWD) which, without any therapy, will end lethally in 15% of all cases. With adequate medical and other interventions lethality is about two percent (Diener, 2003; Wright, Myrick, Henderson, Peters, & Malcolm, 2006). Additionally, the occurrence of an AWS and / or AWD represents a threatening, time-intensive and complex situation for family members (Repper-DeLisi et al., 2008; Yu et al., 2012).

Since 2011, in addition to patients undergoing short-term surgery, also patients with oncological diagnoses are hospitalized in the ENT and Jaw Surgery Department at the University Hospital Basel (USB). These patients are in need of prolonged surgical treatments and resulting longer periods of abstinence from food and drink, including alcohol and other substances, increase the risk of alcohol withdrawal. For instance, in the ENT and Jaw Surgery Department, in 2011, 74 out of 910 inpatients were at risk for or already experienced an AWD and 47 of them needed permanent supervision to guarantee their safety. Bridging the period of abstinence by drinking alcohol pre- and postoperatively is a suboptimal option for these patients due to the relatively long surgical treatment. This situation called for action: based on positive experiences within the dementia-delirium-programme of USB (Hasemann & Pretto, 2006), an evidence-based approach to screen for, detect and treat AWS and / or AWD in ENT and jaw surgery patients was developed and implemented (Hasemann, 2013). Now, this new approach needs to be evaluated.

DETAILED DESCRIPTION:
The aims of the proposed study are to describe patient trajectories and to evaluate the processes and structures of the nurse-led approach in the ENT and Jaw Surgery Department at USB. The following research questions were generated:

Aim 1): Who are the patients captured with the algorithm, what are their risk factors, and how are the patient trajectories in terms of decisions, development, start, duration and ending of AWS and / or AWD? Specific questions asked:

* Which are demographic and medical characteristics of patients?
* How many patients are at risk for AWD / AWS?
* Which decisions do patients make?
* What is the time of onset, duration and ending of AWS and / or AWD?
* Were additional resources used to guarantee safety of patients?

Aim 2): How is the prevention algorithm adhered to? Specific questions asked:

* How many patients were risk-assessed by a nurse at hospital admission?
* How many patients or those who should have been asked were eventually asked to agree to substitution therapy?
* How many patients at risk were assessed using the Clinical Institute Withdrawal Assessment (CIWA)-Ar?
* How many times was the delirium expert consultation service contacted due to reasons stated in algorithm?

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (18 years and older)
* Patient hospitalized with an ENT or jaw carcinoma with required hospitalization for 72 hours and beyond.

Exclusion Criteria:

* non Swiss German speaking patient
* patient being deaf in both ears
* patients with known dementia in history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient hospitalized with an ENT or jaw carcinoma
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Nurses' and doctors' adherence to the patients' surveillance algorithm | baseline until hospital discharge; hospital stay will last 72 hours minimum over a retrospective period of two years
  Percentage of fulfilled steps of the algorithm

SECONDARY OUTCOMES:
Percentage of patients developping alcohol withdrawal delirium under surveillance algorithm | baseline until hospital discharge over a retrospective period of two years; hospital stay will last 72 hours minimum
  Percentage of patients in the substitution programme developping withdrawal delirium

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hasemann, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland

REFERENCES:
- [Background] Bleich S, Sperling W, Wiltfang J, Maler JM, Kornhuber J. [Excitatory neurotransmission in alcoholism]. Fortschr Neurol Psychiatr. 2003 Jul;71 Suppl 1:S36-44. doi: 10.1055/s-2003-40504. German. PMID 12947542
- [Background] Corfee FA. Alcohol withdrawal in the critical care unit. Aust Crit Care. 2011 May;24(2):110-6. doi: 10.1016/j.aucc.2010.08.005. Epub 2010 Sep 25. PMID 20870419
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Foy A, Kay J, Taylor A. The course of alcohol withdrawal in a general hospital. QJM. 1997 Apr;90(4):253-61. doi: 10.1093/qjmed/90.4.253. PMID 9307759
- [Background] Galvin R, Brathen G, Ivashynka A, Hillbom M, Tanasescu R, Leone MA; EFNS. EFNS guidelines for diagnosis, therapy and prevention of Wernicke encephalopathy. Eur J Neurol. 2010 Dec;17(12):1408-18. doi: 10.1111/j.1468-1331.2010.03153.x. PMID 20642790
- [Background] Kuo YR, Jeng SF, Lin KM, Hou SJ, Su CY, Chien CY, Hsueh KL, Huang EY. Microsurgical tissue transfers for head and neck reconstruction in patients with alcohol-induced mental disorder. Ann Surg Oncol. 2008 Jan;15(1):371-7. doi: 10.1245/s10434-007-9506-5. Epub 2007 Nov 1. PMID 17973172
- [Background] Mayo-Smith MF, Beecher LH, Fischer TL, Gorelick DA, Guillaume JL, Hill A, Jara G, Kasser C, Melbourne J; Working Group on the Management of Alcohol Withdrawal Delirium, Practice Guidelines Committee, American Society of Addiction Medicine. Management of alcohol withdrawal delirium. An evidence-based practice guideline. Arch Intern Med. 2004 Jul 12;164(13):1405-12. doi: 10.1001/archinte.164.13.1405. PMID 15249349
- [Background] Nagel M, Ferbert A. [Diseases due to alcoholism]. Fortschr Neurol Psychiatr. 2005 Aug;73(8):470-82; quiz 483-4. doi: 10.1055/s-2004-830191. No abstract available. German. PMID 16052441
- [Background] National Clinical Guideline Centre (UK). Alcohol Use Disorders: Diagnosis and Clinical Management of Alcohol-Related Physical Complications [Internet]. London: Royal College of Physicians (UK); 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK65576/ PMID 22876380
- [Background] Neyman KM, Gourin CG, Terris DJ. Alcohol withdrawal prophylaxis in patients undergoing surgical treatment of head and neck squamous cell carcinoma. Laryngoscope. 2005 May;115(5):786-90. doi: 10.1097/01.MLG.0000160085.98289.E8. PMID 15867640
- [Result] Allen NE, Beral V, Casabonne D, Kan SW, Reeves GK, Brown A, Green J; Million Women Study Collaborators. Moderate alcohol intake and cancer incidence in women. J Natl Cancer Inst. 2009 Mar 4;101(5):296-305. doi: 10.1093/jnci/djn514. Epub 2009 Feb 24. PMID 19244173
- [Result] Awissi DK, Lebrun G, Coursin DB, Riker RR, Skrobik Y. Alcohol withdrawal and delirium tremens in the critically ill: a systematic review and commentary. Intensive Care Med. 2013 Jan;39(1):16-30. doi: 10.1007/s00134-012-2758-y. Epub 2012 Nov 27. PMID 23184039
- [Result] Becker U, Deis A, Sorensen TI, Gronbaek M, Borch-Johnsen K, Muller CF, Schnohr P, Jensen G. Prediction of risk of liver disease by alcohol intake, sex, and age: a prospective population study. Hepatology. 1996 May;23(5):1025-9. doi: 10.1002/hep.510230513. PMID 8621128
- [Result] Delgado-Rodriguez M, Gomez-Ortega A, Mariscal-Ortiz M, Palma-Perez S, Sillero-Arenas M. Alcohol drinking as a predictor of intensive care and hospital mortality in general surgery: a prospective study. Addiction. 2003 May;98(5):611-6. doi: 10.1046/j.1360-0443.2003.00353.x. PMID 12751978
- [Result] Genther DJ, Gourin CG. The effect of alcohol abuse and alcohol withdrawal on short-term outcomes and cost of care after head and neck cancer surgery. Laryngoscope. 2012 Aug;122(8):1739-47. doi: 10.1002/lary.23348. Epub 2012 May 7. PMID 22566069
- [Result] Kraemer KL, Mayo-Smith MF, Calkins DR. Independent clinical correlates of severe alcohol withdrawal. Subst Abus. 2003 Dec;24(4):197-209. doi: 10.1023/a:1026099426602. PMID 14574086
- [Result] O'Brien JM Jr, Lu B, Ali NA, Martin GS, Aberegg SK, Marsh CB, Lemeshow S, Douglas IS. Alcohol dependence is independently associated with sepsis, septic shock, and hospital mortality among adult intensive care unit patients. Crit Care Med. 2007 Feb;35(2):345-50. doi: 10.1097/01.CCM.0000254340.91644.B2. PMID 17205003
- [Result] Repper-DeLisi J, Stern TA, Mitchell M, Lussier-Cushing M, Lakatos B, Fricchione GL, Quinlan J, Kane M, Berube R, Blais M, Capasso V, Pathan F, Karson A, Bierer M. Successful implementation of an alcohol-withdrawal pathway in a general hospital. Psychosomatics. 2008 Jul-Aug;49(4):292-9. doi: 10.1176/appi.psy.49.4.292. PMID 18621934
- [Result] Spies CD, Dubisz N, Funk W, Blum S, Muller C, Rommelspacher H, Brummer G, Specht M, Hannemann L, Striebel HW, et al. Prophylaxis of alcohol withdrawal syndrome in alcohol-dependent patients admitted to the intensive care unit after tumour resection. Br J Anaesth. 1995 Dec;75(6):734-9. doi: 10.1093/bja/75.6.734. PMID 8672322
- [Result] Yu YH, Chen AC, Hu CC, Hsieh PH, Ueng SW, Lee MS. Acute delirium and poor compliance in total hip arthroplasty patients with substance abuse disorders. J Arthroplasty. 2012 Sep;27(8):1526-9. doi: 10.1016/j.arth.2011.12.003. Epub 2012 Feb 8. PMID 22325962